CLINICAL TRIAL: NCT00699413
Title: Supplements for Controlling Resistance to Insulin
Acronym: SCORE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decided to withdraw from study.
Sponsor: University of Southern California (Other)
Collaborators: InterHealth Nutraceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Michael I. Goran, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCORE1
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - nutrition education plus active supplement (Active Comparator): nutrition education plus active supplement
  Interventions: Drug: nutrition education plus active supplement
- 2 - nutrition education plus inactive supplement (Placebo Comparator): nutrition education plus inactive supplement
  Interventions: Drug: nutrition education plus inactive supplement

INTERVENTIONS:
Drug: nutrition education plus active supplement — After all baseline measures have been completed, participants will be randomly assigned to either the nutrition education + supplement group, or the nutrition education + placebo group. The length of the intervention is twelve weeks. Nutrition classes will take place once a week for 1 1/2 hours. Subjects will be encouraged to increase fiber and decrease sugar intake. They will also be separated into gender-specific classes.
  Active and inactive supplements will be identical in appearance and taste. Active supplements will contain 2,700 mgs/day of Super CitriMax (hydroxycitrate)and 400 µg per day of ChromeMate (niacin-bound Chromium). Supplements will be in powder and tablet form, and should be taken 30 minutes prior to each meal.
  Other Names: none known
  Arms: 1 - nutrition education plus active supplement
Drug: nutrition education plus inactive supplement — After all baseline measures have been completed, participants will be randomly assigned to either the nutrition education + supplement group, or the nutrition education + placebo group. The length of the intervention is twelve weeks. Nutrition classes will take place once a week for 1 1/2 hours. Subjects will be encouraged to increase fiber and decrease sugar intake. They will also be separated into gender-specific classes.
  Active and inactive supplements will be identical in appearance and taste.
  Other Names: none known
  Arms: 2 - nutrition education plus inactive supplement

SUMMARY:
The purpose of this study is to evaluate the effects of a combination of hydroxcycitrate (HCA) and niacin-bound chromium, in conjunction with nutrition education, over a twelve week period. Participants will be evaluated with regard to BMI, percent body fat, insulin activity, and hunger.

DETAILED DESCRIPTION:
The prevalence of obesity among youth has increased dramatically in recent years. Parallel to the increased rates of pediatric obesity, overweight children present clinically with adiposity related comorbidities such as insulin resistance and type 2 diabetes. The prevailing recommendations for overweight youth are to increase physical activity levels and limit energy intake in order to improve body composition. Currently there is little empirical evidence to support the efficacy of these recommendations. Alternatively, evidence in adults suggests that nutritional supplementation with (-) hydroxycitric acid (HCA), an organic acid found naturally in citrus fruits, and chromium may lead to favorable changes in body composition and improve glucose regulation. To date, these issues have not been tested in youth. Therefore, the purpose of the present investigation is to examine the effects of a nutritional education program combined with either HCA + chromium or placebo on measures of body composition and glucose regulation in overweight adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age

  * All subjects will be between 13 and 17 years of age
* Overweight

  * All subjects will be overweight as defined by an age & sex-specific body mass index ≥ 85th percentile based on CDC BMI growth charts [US Department of Health and Human Services, 2000], calculated by Epi Info Software, version 3.3.

Exclusion Criteria:

* Presently taking any prescribed medication(s) or diagnosed with any syndrome or disease that could influence dietary intake, body composition and fat distribution, or insulin action or secretion.
* Previously diagnosed with any major illness since birth (e.g. sever intrauterine growth retardation, chronic birth asphyxia, cancer).
* Children with type 1 and/or type 2 diabetes will be excluded are referred to a physician.
* Currently involved with any dietary, exercise, or weight loss program or have been in the 6 months prior to participation.
* Unexplained weight loss or gain in the prior six months.
* Oral contraception use in sexually active females
* Children who live further than 20 miles away from the USC Health Science Campus (HSC).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC - Preventive Medicine, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: nutrition education plus active supplement
- Control Arm: nutrition education plus inactive supplement
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 4 | 4
Completed | 0 | 0
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Study terminated by sponsor | 4 | 2

BASELINE CHARACTERISTICS:
Population: * Two control participants withdrew prior to data collection.
  * Study terminated prior to complete data collection of remaining participants (only partial data presented in results section).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.41) | 14 (1) | 14.6 (1.37)
Age, Customized [Number; unit: participants]
  <=18 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index
Description: Change in Body Mass Index measurement at baseline and 12 weeks
Time Frame: measured at baseline and 12 weeks
Population: Data were not collected. Previously reported data were incorrect and do not reflect a change in BMI from baseline to 12 weeks. Only basic demographic information was collected at baseline and no outcome measures were captured. The study was terminated prior to the 12 week intervention end and no data were collected at the second time point.
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Insulin Activity
Description: Change in insulin activity measured at baseline and 12 weeks
Time Frame: Measured at baseline and 12 weeks
Population: Data were not collected
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Body Fat
Description: Change in percent body fat measured at baseline and 12 weeks
Time Frame: Measured at baseline and 12 weeks
Population: Data were not collected
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hunger
Description: Change in hunger score using Likert scale measured at baseline and 12 weeks
Time Frame: Measured at baseline and 12 weeks
Population: Data were not collected
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intervention Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No